CLINICAL TRIAL: NCT06131931
Title: Connecting Latinos En Pareja: a Couples-based HIV Prevention Intervention for Latino Male Couples
Brief Title: HIV Prevention Intervention for Latino Male Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005650; 1R01MD018963-01A1 (NIH)
Record Dates: First submitted 2023-11-04; First posted 2023-11-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: HIV
Keywords: HIV; Latino; male; couples

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connecting Latinxs en Pareja (CLP) (Experimental): CLP is a four-session intervention grounded in social cognitive theory and a relationship oriented ecological framework.
  Interventions: Other: CLP Intervention
- Wellness Promotion (WP) (Active Comparator): WP focuses on nutrition, fitness, healthcare, and stress management and emphasizes adherence to medical regimens and medication management.
  Interventions: Other: WP Intervention

INTERVENTIONS:
Other: CLP Intervention — 4 weekly sessions lasting approximately 60 minutes that will be audio recorded for quality assurance. Each couple will be assigned one RA who will serve as their facilitator and guide them through the Connecting Latinxs en Pareja (CLP) sessions. The RA will deliver the appropriate intervention in either Spanish or English at the couple's preference. Sessions will be delivered via zoom (or comparable secure platform), using established procedures from the team's prior studies. Each participant will complete Qualtrics assessments at baseline, 3-, 6- and 9-months post randomization and biological (hair biomarkers for PrEP and ART adherence) and behavioral and psychosocial data collected.
  Arms: Connecting Latinxs en Pareja (CLP)
Other: WP Intervention — 4 weekly sessions lasting approximately 60 minutes that will be audio recorded for quality assurance. Each couple will be assigned one RA who will serve as their facilitator and guide them through the Wellness Promotion (WP) sessions. The RA will deliver the appropriate intervention in either Spanish or English at the couple's preference. Sessions will be delivered via zoom (or comparable secure platform), using established procedures from the team's prior studies. Each participant will complete Qualtrics assessments at baseline, 3-, 6- and 9-months post randomization and biological (hair biomarkers for PrEP and ART adherence) and behavioral and psychosocial data collected.
  Arms: Wellness Promotion (WP)

SUMMARY:
The primary objective of this proposal is to test the efficacy of Connecting Latinxs en Pareja (CLP). CLP is a four-session intervention grounded in social cognitive theory and a relationship oriented ecological framework.

The investigators will examine whether participants assigned to CLP report an increase in the proportion of HIV protected anal sex acts to those assigned to a Wellness Promotion (WP) time and attention matched control condition. The primary outcome, relates to use of HIV protection.

DETAILED DESCRIPTION:
The investigators will recruit 200 Latinx male couples (N=400 individuals) from 50 Ending the HIV Epidemic (EHE) jurisdictions and an additional 17 areas with high HIV burden among Latinxs. Building from our previous success in engaging sexual minority Latinx men, the investigators will implement a multipronged recruitment strategy, including social media and social networking apps and venue-based recruitment. Couples will be randomly assigned to CLP or a piloted Wellness Promotion (WP) time and attention matched control condition. Follow- up will occur every 3 months over 9 months, and biological (hair biomarkers for Pre-Exposure Prophylaxis (PrEP) and Antiretroviral Therapy (ART) adherence) and behavioral and psychosocial data collected. The primary outcome, HIV protection, is operationalized with a validated composite algorithm as protected acts of anal intercourse (i.e., anal sex acts in which condoms, PrEP, or Treatment as Prevention (TasP) are used to reduce risk of HIV transmission) within the couple and with outside partners. Guided by the Designing for Dissemination and Sustainability (D4DS) framework, the investigators will derive practical recommendations and considerations for sustainability and scaling up of the intervention (or other next steps). All intervention sessions will be conducted via Zoom by a facilitator. The facilitator will conduct all remote sessions from a private office at the University of Central Florida College of Medicine. Study participants will collect their own hair samples and mail it back to the University of California San Francisco. Participants will receive the collection toolkit and paid stamped mail package to ship samples. Hair sample collection is noninvasive and does not require specific skills, sterile equipment, or specialized storage. Samples can be stored at room temperature for long periods prior to analysis and shipped without taking the precautions associated with biohazardous materials.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* reside in the 50 local jurisdictions identified by the EHE initiative or 17 jurisdictions with most HIV diagnoses among Latinxs
* identify as Latinx/Hispanic/Afro-Latinx or reports having a main partner who identifies as Latinx/Hispanic/Afro-Latin
* report having a main/primary male partner operationalized as a man with whom he has a primary ongoing sexual relationship, for at least 3 months
* at least one member of the dyad report three acts of unprotected of anal sex (with main or other partners)
* able to speak English and/or Spanish

Exclusion Criteria:

Either partner:

* reports severe intimate partner violence (IPV) within the dyad during the past year on the Revised Conflict Tactic Scale[1-4]
* has a language or cognitive impairment that would prevent informed consent. Inclusion of dyads reporting severe IPV could pose dangers and ethical concerns and will be referred to domestic abuse organizations for screening and services.
* adults unable to consent
* pregnant women
* prisoners
* individuals who are not yet adults

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Latinx men and their same-sex partners
Enrollment: 400 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
HIV Prevention sessions and assessments | 4 years
  The investigators will examine whether participants assigned to CLP report an increase in the proportion of HIV protected anal sex acts to those assigned to a Wellness Promotion (WP) time and attention matched control condition by conducting weekly sessions and assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No